CLINICAL TRIAL: NCT03504345
Title: Assessing the Optimal Duration of Progesterone Supplementation Prior to Transfer of Frozen Embryos in the Recurrent Implantation Failure Population
Brief Title: Progesterone Supplementation in Frozen Embryo Transfer Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Crystal Chan, Clinician Investigator, Assistant Professor, Department of Obstetrics & Gynaecology, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Infertility Due to Nonimplantation; Infertility
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This arm of the study will have their frozen-thawed embryo transfer take place on the sixth day of progesterone supplementation (Prometrium), which is the standard protocol in our clinic.
  Interventions: Drug: Prometrium
- Experimental Group (Experimental): This arm of the study will have their frozen-thawed embryo transfer take place on the seventh day of progesterone supplementation (Prometrium).
  Interventions: Drug: Prometrium

INTERVENTIONS:
Drug: Prometrium — The intervention will involve delaying the transfer of a frozen-thawed embryo into the uterus to increase the duration of progesterone exposure.

SUMMARY:
Recurrent implantation failure (RIF) occurs after women undergo in vitro fertilization and have multiple embryos transferred but no resulting pregnancies. RIF is a very challenging clinical entity for the reproductive physician and the patient. In fact, there is not even an agreed upon definition in the medical community. Many potential causes have been investigated over the past several years but no clear answer has emerged. Interest has recently turned to the endometrium, or the lining of the uterus. Studies have shown that the genes that are turned on in the endometrium vary based on how long this tissue has been exposed to progesterone, an important hormone that prepares the uterine lining for implantation of the growing embryo. In some women, it seems that they require longer periods of progesterone exposure to reach the same state of readiness. We hypothesize that an even larger proportion of women in RIF population will require longer treatments with progesterone.

In this study, we will randomize women with RIF who are about to undergo a frozen embryo transfer to one of two groups. The first group will have their embryo transfer done on the standard sixth day of progesterone treatment. The other group will have their transfer done on the seventh day of progesterone. We will be comparing the clinical pregnancy rate of the two groups as well as the live birth rate and miscarriage rate. We expect that extending the progesterone treatment by one day will increase the pregnancy rate of women with RIF.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Mount Sinai Fertility who wants to undertake a frozen embryo transfer
* History of recurrent implantation failure, defined as no pregnancy after three or more embryo transfers of four or more good quality blastocysts

Exclusion Criteria:

* Previous testing with Endometrial Receptivity Assay (ERA)
* Unable understand/communicate in English

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 6 to 8 weeks after embryo transfer
  Rate of pregnancy, evidenced by clinical (fetal heartbeat) or ultrasound parameters (ultrasound visualization of a gestational sac, embryonic pole with heartbeat). It includes ectopic pregnancy.

SECONDARY OUTCOMES:
Live birth rate | Approximately 9 months after embryo transfer
  Rate of birth in which a fetus is delivered with signs of life after complete expulsion or extraction from its mother, beyond 20 completed weeks of gestational age
Miscarriage rate | Approximately 3 months after embryo transfer
  Rate of natural death of embryo or fetus, after reaching clinical pregnancy stage and at or before 10 weeks gestation.

IPD SHARING:
Plan to Share IPD: No